CLINICAL TRIAL: NCT03884257
Title: A Randomized Controlled Non-inferiority Trial to Evaluate the Safety and Efficacy of the Passeo-18 Lux Drug-coated Balloon of Biotronik in the Treatment of Subjects with Stenotic, Restenotic or Occlusive Lesions of the Femoropopliteal Artery Compared to the Medtronic IN.PACT Admiral Drug-coated Balloon
Brief Title: A Trial to Evaluate the Safety and Efficacy of the Passeo-18 Lux Drug-coated Balloon of Biotronik in the Treatment of the Femoropopliteal Artery Compared to the Medtronic IN.PACT Admiral Drug-coated Balloon.
Acronym: BIOPACT-RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ID3 Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIOPACT-RCT_V1.0_14DEC2018
Record Dates: First submitted 2019-03-11; First posted 2019-03-21 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: The patients will be assigned at random to one of two treatment groups namely the Passeo-18 Lux or the IN.PACT Admiral treatment group.
Who Masked: Participant
Masking Description: a single-blind masking will be implemented. The patient won't know which DCB he/she received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passeo-18 Lux treatment group (Experimental): These patients will be treated with the Passeo-18 Lux (Biotronik).
  Interventions: Device: Passeo-18 Lux treatment group
- IN.PACT Admiral treatment group (Active Comparator): These patients will be treated with the IN.PACT Admiral (Medtronic).
  Interventions: Device: IN.PACT Admiral treatment group

INTERVENTIONS:
Device: Passeo-18 Lux treatment group — Percutaneous endovascular angioplasty with the Passeo-18 lux
  Arms: Passeo-18 Lux treatment group
Device: IN.PACT Admiral treatment group — Percutaneous endovascular angioplasty with the IN.PACT Admiral
  Arms: IN.PACT Admiral treatment group

SUMMARY:
The BIOPACT RCT tiral investigates the efficacy and safety of stenosis, restenosis or occlusions in the femoropopliteal artery of patients presenting a rutherford classification 2,3 or 4 with a Passeo-18 Lux drug-coated balloon of Biotronik. The Paclitaxel eluting balloons are designed for percutaneous transluminal angioplasties in which the balloon will dilate the artery upon inflation and deliver the paclitaxel locally.

An expected total of 151 patients will be treated with the Passeo-18 Lux and compared to a control group of another 151 patients that will be treated with the IN.PACT Admiral drug-coated balloon of Medtronic. Assignment to the treatment groups will be at random. The study will be conducted in two phases. A first pilot study phase of 120 patients distributed evenly over both treatment groups and a second phase to formally test the non-inferiority hypothesis.

The balloon is coated with Paclitaxel intended to avoid cellular proliferation. The drug is released by means of rapid inflation as to release a high dose in a short amount of time. Patients will be invited for a follow-up visit at 1, 6 and 12 months post-procedure.

The primary efficacy endpoints are defined as follows. Freedom from clinically-driven target lesion revascularization at 12 months. Freedom from device- and procedure-related death through 30 days post-index procedure, major target limb amputation through 12 months post-procedure and clinically-driven target vessel revascularization through 12 months post-index procedure. The secondary endpoints are defined as acute device success, acute procedural success , freedom from all cause of death, major target limb amputation and clinically driven target vessel revascularisation through 30 days post-procedure, sustained clinical improvement, no major adverse events through 6 and 12 months post-procedure, primary patency, target lesion revascularisation, target vessel revascularisation, binary restenosis, major target limb amputation, thrombosis at target lesion, change of walking impairment questionnaire score from baseline, change in target limb rutherford classification or ABI.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to assess the safety and efficacy of the Passeo-18 Lux DCB for the treatment of stenotic, restenotic or occlusive lesions of the femoropopliteal arteries. Furthermore a non-inferiority hypothesis will be tested with the IN.PACT Admiral DCB as comparator.

The patients will be selected based on the investigator's assessment, evaluation of the underlying disease and the eligibility criteria. The patient's medical condition should be stable, with no underlying medical condition which would prevent them from performing the required testing or from completing the study. Patients should be geographically stable, willing and able to cooperate in this clinical study, and remain available for long term follow-up. The patient is considered enrolled in the study after obtaining the patients informed consent, if there is full compliance with the study eligibility criteria and after successful guidewire passage through the study target lesion.

Prior to the index procedure the following will be collected: an informed consent for data collection, demographics, medical history, medication record, physical examination, clinical category of acute limb ischemia (Rutherford category), the resting ankle-brachial index (ABI), blood sample test (complete blood count, comprehensive metabolic panel and if applicable pregnancy test) and a walking impairment questionnaire.

During the procedure the guidewire will cross the entire study lesion after which the lesion will be assessed through angiography. A pre-dilatation with a standard non-drug-coated balloon will be performed followed by a dilatation of the lesion with either a Passeo-18 Lux (Biotronik) or an IN.PACT Admiral balloon (Medtronic). If dilatation was not successful (>30% stenosis, perforation, occlusive or flow limiting dissection) prolonged inflation should be attempted after which bail-out stenting with a bare nitinol stent is allowed in case of inadequate results.

The regular follow-up is necessary to monitor the condition of the patient and the results of the procedure. The patients will be invited for the following required follow-up visits at 1,6 and 12 months. During these visit the following data will be collected: medication record, physical exam, target limb ABI and Rutherford classification, duplex ultrasound of target vessel, walking impairment questionnaire and possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years
* Subject has Rutherford classification 2, 3 or 4
* Subject has provided written informed consent and is willing to comply with study follow- up requirements
* De novo stenotic or occlusive lesion(s) or non-stented restenotic or occlusive lesion(s) occurring >90 days after prior plain old balloon (POBA) angioplasty or >180 days after prior DCB treatment
* Target lesion is located between the ostium of the SFA and the end of the P1 segment of the popliteal artery
* Target vessel diameter ≥4mm and ≤7mm
* Target lesion must be stenotic lesion ≤180mm in length (one long lesion or tandem lesions) by investigator's visual estimate or a total occlusion ≤120mm in length by investigator's visual estimate.

Note: tandem lesions must have a total length of ≤180mm by visual estimate and be separated by ≤30mm

* Target lesion must have angiographic evidence of ≥70% stenosis by investigator's visual estimation
* Successful, uncomplicated crossing of the target lesion occurs when the tip of the guide wire is distal to the target lesion without the occurrence of flow-limiting dissection or perforation and is judged by visual inspection to be within the true lumen. Subintimal dissection techniques may be used if re-entry occurs above the knee (ATK) and without the use of re-entry devices
* Target lesion is located at least 30mm from any stent, if target vessel was previously stented
* After pre-dilatation, the target lesion is ≤50% residual stenosis, absence of a flow-limiting dissection and treatable with available device matrix
* A patent inflow artery free from significant stenosis (≥50% stenosis) as confirmed by angiography
* At least one patent native outflow artery to the ankle or foot, free from significant stenosis (≥50% stenosis) as confirmed by angiography

Exclusion Criteria:

* Acute limb ischemia
* Patient underwent an intervention involving the target vessel within the previous 90 days
* Patient underwent any lower extremity percutaneous treatment in the ipsilateral limb using a paclitaxel-eluting stent or DCB within the previous 90 days
* Patient underwent a percutaneous transluminal angioplasty (PTA) of the target lesion using a DCB within the previous 180 days
* Women who are pregnant, breast-feeding or intend to become pregnant
* Patient has life expectancy of less than 1 year
* Patient has a known allergy to contrast medium that cannot be adequately pre-medicated
* Patient is allergic to all antiplatelet treatments
* Patient is receiving immunosuppressant therapy
* Patient has platelet count <100.000/mm3 or >700.000/mm3
* Patient has history of gastrointestinal haemorrhage requiring a transfusion within 3 months prior to the study procedure
* Patient is diagnosed with coagulopathy that precludes treatment with systemic anticoagulation and/or dual antiplatelet therapy (DAPT)
* Patient has history of stroke within the past 90 days
* Patient has history of myocardial infarction within the past 30 days
* Patient is participating in an investigational drug or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints from this study, or patient is planning to participate in such study prior to the completion of this study
* Patient has had any major (e.g. cardiac, peripheral, abdominal) surgical procedure or intervention unrelated to this study within 30 days prior to the index procedure or has planned major surgical procedure or intervention within 30 days of the index procedure
* An intervention in the contralateral limb, planned within 30 days post-index procedure
* Patient had previous bypass surgery of the target lesion
* Patient had previous treatment of the target vessel with thrombolysis or surgery
* Patient is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol
* Target lesion involves an aneurysm or is adjacent to an aneurysm (within 5mm)
* Target lesion requires treatment with alternative therapy such as stenting, laser, atherectomy, cryoplasty, brachytherapy or re-entry devices
* Significant target vessel tortuosity or other parameters prohibiting access to the target lesion
* Presence of thrombus in the target vessel
* Iliac inflow disease requiring treatment, unless the iliac artery disease is successfully treated first during the index procedure. Success is defined as ≤30% residual diameter stenosis without death or major complications
* Presence of an aortic, iliac or femoral artificial graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
freedom from clinically-driven target lesion revascularization (CD-TLR) at 12 months post-procedure | 12 months post-procedure
  defined as any reintervention at the target lesion due to the following symptoms: drop of ABI >20% or ABI >0.15 compared to the post-procedure ABI.
Safety composite: number of participants who deceased, had major amputation, or target vessel revascularization (CD-TVR) | 12 months post-procedure
  composite of (1) freedom from device- and procedure-related death through 30 days post-index procedure, (2) freedom from major target limb amputation (above-the-ankle (ATA)) through 12 months post-procedure or (3) clinically-driven target vessel revascularization (CD-TVR) through 12 months post-index procedure

SECONDARY OUTCOMES:
acute device success | Index procedure
  defined as successful delivery, balloon inflation, deflation and retrieval of the intact study device without burst below rated burst pressure
acute procedural success | index procedure
  defined as restoration of the target lesion with ≤30% residual stenosis in the final angiogram
freedom from all causes of death, freedom from major target limb amputation and freedom from CD-TVR through 30 days | 1 month post-procedure
  freedom from all cause death, major target limb amputation and CD-TVR through 30 days post-procedure
Sustained clinical improvement | 6 and 12 months post-procedure
  defined as freedom from major target limb amputation, TVR, worsening target limb Rutherford class (compared to baseline) and decrease in target limb ankle brachial index (ABI) or toe brachial index (TBI) ≥0.15 (compared to baseline)
freedom from major adverse events | 6 and 12 months post-procedure
  defined as composite of all-cause death, CD-TVR and major target limb amputation, or thrombosis at the target lesion
primary patency rate | 6 and 12 months post-procedure
  defined as a composite of freedom from clinically-driven target lesion revascularization (CD-TLR) and binary restenosis (restenosis defined as duplex ultrasound (DUS) peak systolic velocity ratio (PSVR) ≥2.4 or ≥50% stenosis as assessed by an independent DUS core lab) through 12 months post-index procedure
freedom from target lesion revascularisation | 6 and 12 months post-procedure
  defined as a reintervention to maintain or restore the patency in the target lesion. TLR is clinically-driven (CD) when the TLR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure
freedom from target vessel revascularisation | 6 and 12 months post-procedure
  defined as a reintervention to maintain or restore the patency in the target vessel. TVR is clinically-driven (CD) when the TVR was needed due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure
freedom from binary restenosis | 6 and 12 months post-procedure
  defined as restenosis confirmed by DUS PSVR ≥2.4 or ≥50% stenosis as assessed by independent angiographic and DUS core labs
freedom from major target limb amputation | 6 and 12 months post-procedure
  defined as an amputation above the ankle in the target limb
freedom from thrombosis at target lesion | 6 and 12 months post-procedure
  freedom from thrombosis at target lesion
change in walking impairment questionnaire score from baseline to 6 and 12 months | 6 and 12 months post-procedure
  change in walking impairment questionnaire (WIQ) score from baseline to 6 and 12 months.
  The WIQ consists of 6 sections each consisting of multiple questions. Each question is scored from 0 to 4 (0 meaning a lot of problems and 4 no problems at all). The scores per section are summed up and recalculated to percentages (100% meaning very good and 0% meaning very bad). All the sections are averaged to give the final WIQ-score.
change in target limb rutherford class from baseline to 6 and 12 months | 6 and 12 months post-procedure
  change in target limb rutherford class from baseline to 6 and 12 months
change in target limb resting ABI or TBI from baseline to 6 and 12 months | 6 and 12 months post-procedure
  change in target limb resting ABI or TBI from baseline to 6 and 12 months
freedom from all causes of death | 6 and 12 months post-procedure
  freedom from all causes of death

CONTACTS AND LOCATIONS:
Overall Officials: Koen Deloose, MD, Principal Investigator — AZ Sint-Blasius
Locations (14):
- Austria (2):
  - Medical University of Graz, Graz, Graz
  - Hanusch Hospital, Vienna, Vienna
- Belgium (6):
  - UZA, Antwerp, Antwerp
  - OLV Ziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
  - Z.O.L., Genk
  - R.Z. Heilig Hart, Tienen
- France (4):
  - CHU Bordeaux, Bordeaux, Nouvelle-Aquitaine
  - Clinique Pasteur, Toulouse, Occitanie
  - Clinique Rhône Durance, Avignon, Provence-Alpes-Côte d'Azur Region
  - Hopital Paris Saint Joseph, Paris
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Triemlispital Zürich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deloose K, Lansink W, Brodmann M, Werner M, Keirse K, Goueffic Y, Verbist J, Maene L, Hendriks J, Brunet J, Ducasse E, Levent K, Sauguet A, Deglise S, Vandael F. Methodology of the BIOPACT RCT, a Multi-center, Randomized, Non-inferiority Trial Evaluating Safety and Efficacy of Passeo-18 Lux Drug-Coated Balloon (DCB) of Biotronik Compared to the Medtronic IN.PACT Admiral DCB in the Treatment of Subjects with Lesions of the Femoropopliteal Artery. Cardiovasc Intervent Radiol. 2022 Dec;45(12):1855-1859. doi: 10.1007/s00270-022-03259-z. Epub 2022 Sep 4. PMID 36058996